CLINICAL TRIAL: NCT03938571
Title: Torsby I Trial: A Prospectively Randomized Study on Standard Duodenal Switch vs. Single Anastomosis Duodeno-ileostomy Duodenal Switch
Brief Title: Standard Duodenal Switch vs. Single Anastomosis Duodeno-Ileostomy Duodenal Switch
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Värmland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/133
Record Dates: First submitted 2019-03-11; First posted 2019-05-06 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Obesity; Surgery; Metabolic Syndrome; Malnutrition
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard DS (Experimental): Standard duodenal switch:
  1. Sleeve gastrectomy over a 35 Fr bougie
  2. Division of the duodenum 2-3 cm distally of the pylorus
  3. Measurement of the small bowel. 100 cm common channel. 150 cm alimentary limb.
  4. Duodenoileostomy completely handsewn with 250 cm distance to the ileocecal valve.
  5. Entero-entero-anastomosis linear stapled and handsewn.
  6. Division between the two anastomosis.
  7. Closure of the mesenteric defects.
  Interventions: Procedure: Duodenal Switch
- SADI-DS (Active Comparator): Duodenal switch with Single anastomosis duodeno-ileostomy:
  1. Sleeve gastrectomy over a 35 Fr bougie
  2. Division of the duodenum 2-3 cm distally of the pylorus
  3. Measurement of the small bowel. 250 cm alimentary limb/common channel.
  4. Duodenoileostomy completely handsewn with 250 cm distance to the ileocecal valve.
  5. Closure of the mesenteric defects.
  Interventions: Procedure: Duodenal Switch

INTERVENTIONS:
Procedure: Duodenal Switch

SUMMARY:
The aim of the Torsby I Trial is to identify differences and similarities between a standard duodenal switch (DS) and a single-anastomosis duodeno-ileostomy (SADI) regarding effect on weight, comorbidities and malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 45
* Ability to understand the legal background of a study

Exclusion Criteria:

* Previous bariatric or anti-reflux surgery
* Drug-abuse
* Inflammatory bowel disease
* Complex psychiatric situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change of weight (kg) | January 2024 (5 yr follow-up) and january 2029 (10 yr follow-up)
  Change of weight in kg with calculation of the relative weight-loss under the follow-up
Early complications | Up to 10 years after operation
  Rate of minor and major complications

SECONDARY OUTCOMES:
Alterations in comorbidities (hypertension) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of the metabolic profile (hypertension).
Alterations in comorbidities (diabetes) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of the metabolic profile (diabetes)
Alterations in comorbidities (sleeping apnea) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of the metabolic profile (sleeping apnea)
Alterations in comorbidities (hyperlipideamia) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of the metabolic profile (hyperlipidemia)
Development of malnutrition (protein) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of levels of protein
Development of malnutrition (vitamin A) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of levels of vitamin A
Development of malnutrition (vitamin D) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of levels of vitamin D
Development of malnutrition (vitamin B12) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of levels of vitamin B12
Development of malnutrition (vitamin B6) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of levels of vitamin B6
Development of malnutrition (vitamin B1) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of levels of vitamin B1
Development of malnutrition (vitamin E) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of levels of vitamin E
Development of malnutrition (calcium) | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Changes of levels of calcium
Late minor complications | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Rate of minor complications (Clavien Dindo < IIIB)
Late major complications | January 2021 (2 yr follow-up), january 2024 (5 yr follow-up), january 2029 (10 yr follow-up)
  Rate of major complications (Clavien Dindo > and = IIIB)

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Hansske, M.D., Study Chair — Consultant

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Axer S, Al-Tai S, Ihle C, Alwan M, Hoffmann L. Perioperative Safety and 1-Year Outcomes of Single-Anastomosis Duodeno-Ileal Bypass (SADI) vs. Biliopancreatic Diversion with Duodenal Switch (BPD/DS): A Randomized Clinical Trial. Obes Surg. 2024 Sep;34(9):3382-3389. doi: 10.1007/s11695-024-07421-z. Epub 2024 Jul 23. PMID 39042310